CLINICAL TRIAL: NCT02038556
Title: Exploring the Outcomes and Financial Impact of a CBT-I Group Program Provided by Registered Nurses for Adults With Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Wendy R. Moore, Registered Nurse, Mayo Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-006921
Record Dates: First submitted 2013-06-10; First posted 2014-01-16 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-05

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cognitive behaviorial therapy for insomnia group program (Experimental): Behavioral
  Interventions: Behavioral: cognitive behaviorial therapy -Insomnia

INTERVENTIONS:
Behavioral: cognitive behaviorial therapy -Insomnia

SUMMARY:
The purpose of this pilot study is to evaluate our RN CBT-I program outcomes and determine utility of this program as a high-value care model targeted specifically to our sleep center patient population.

Hypothesis: PIRS will improve from baseline to 2 month follow up

ELIGIBILITY:
* Able to speak english
* Referred to Mayo Center for Sleep medicine Cognitive behaviorial therapy program for insomnia
* no dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-05; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Pittsburg insomnia rating scale | up to 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Moore, RN, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Mayo Clinic, Rochester, Minnesota